CLINICAL TRIAL: NCT04508647
Title: Ublituximab as Initial Therapy for Treatment-naive Follicular or Marginal Zone Lymphoma With Response-driven Addition of Umbralisib for Suboptimal Response
Brief Title: Ublituximab Followed by Response-driven Addition of Umbralisib for Treatment-naive Follicular or Marginal Zone Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-2128.cc; NCI-2021-00405 (Other: CTRP); U2-NTG-009 (Other: TG Therapeutics Inc.)
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Marginal Zone Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular | interventions — ublituximab; umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ublituximab Only (Experimental): Treatment-Naive Stage II (non-contiguous), Stage III, Stage IV FL + MZL will receive Ublituximab 900mg IV weekly x 4 doses. End of treatment assessment 8 weeks post last dose of single agent ublituximab will be performed.
  Interventions: Drug: Ublituximab
- Ublituximab first, then Ublituximab and Umbralisib (Experimental): Patients who achieve less than a complete response will receive a combination of ublituximab AND umbralisib for a total of 12 cycles. (In the combination arm ublituximab will be administered on day 1,8 and 15 on cycle 1 and on day 1 on each cycle thereafter. Umbralisib will be administered at 800 mg daily for 12 cycles)
  Interventions: Drug: Ublituximab; Drug: Umbralisib

INTERVENTIONS:
Drug: Ublituximab — Ublituximab will be administered as an intravenous infusion through a dedicated line. All infusions will be administered per institutional guidelines.
  During ublituximab monotherapy (initial treatment), Cycle 1 Day 1 administration time frame: Over 4 hours. Cycle 1 days 8 and 15 will be over 3 hours, and Cycle 1 Day 22 will be over 90 minutes. During combination treatment with umbralisib, ublituximab will be administered over 90 minutes.
Drug: Umbralisib — Umbralisib will be administered orally once daily within 30 minutes of starting a meal.
  Arms: Ublituximab first, then Ublituximab and Umbralisib

SUMMARY:
This is an open-label, Phase II interventional study in order to assess efficacy and safety of single agent ublituximab as initial therapy for FL (Follicular lymphoma) and MZL (Marginal zone lymphoma ) with response driven addition of umbralisib for suboptimal response.

DETAILED DESCRIPTION:
Based on overall reporting in low tumor burden FL and MZL, CR rate of at least 30% was achieved when single agent rituximab was used in these subsets. The investigators assume that by administering ublituximab (both as a single agent and in combination with umbralisib for individuals who fail to achieve a CR [Complete response] with the single agent), the CR rate will increase to 50%. Efficacy will be assessed using the proportion of patients treated with ublituximab alone or with ublituximab administered in combination who have a complete response. Thus, the investigators will test the efficacy of ublituximab using a difference in proportions design by comparing an expected study population control rate of 50% to the comparison proportion being determined by the historical control CR rate of 30%. In other words, the null hypothesis is that the true response rate is 30%, and it will be formally tested against a one-sided alternative that the response rate is 50%.

ELIGIBILITY:
Inclusion Criteria:

Disease Related

1. Subjects with histologically documented Follicular lymphoma CD20+ (Grade 1, 2 or 3a) OR Marginal zone lymphoma CD20+ (nodal, extranodal or splenic) according to World Health Organization (WHO) criteria.
2. Ann Arbor Stage II (Non-contiguous), III or IV disease
3. Patients must have a whole body or limited whole body PET/CT scan performed within 42 days prior to registration. CT portion of PET/CT will be done with contrast based on current NCCN guidelines unless patient has borderline renal function or allergic to contrast dye.
4. Patients must have bone marrow biopsy performed within 6 months prior to registration
5. Measurable node must have an LDi greater than 1.5 cms. In the absence of nodal lesions, measurable extranodal disease should have an LDi greated than 1 cm. In patients with Splenic Marginal Zone lymphoma, in the absence of nodal lesions, spleen size should should be over 14 cms with evidence of lymphoma in the bone marrow biopsy.
6. For low tumor burden lymphomas (as determined by GELF criteria) : Include patients diagnosed within 2 years of diagnosis. Low tumor burden patients diagnosed more than 2 years from study entry will be allowed provided patients have documented progression.

Prior Therapy Criteria

1. Patients must be untreated advanced stage disease (Stage III or Stage IV) or Stage II (noncontiguous). (Exception: Involved field or involved site radiation given for localized diagnosis is not considered a line of therapy).

Clinical/Laboratory Criteria

1. Patients must be ≥ 18 years of age and be able to swallow and retain oral medication
2. ECOG performance status of 0-2
3. Patients must have adequate bone marrow function as evidenced by ANC ≥ 1000/µL and platelets ≥ 50,000µL and Hb >= 8g/dl within 28 days prior to registration unsupported by growth factors.
4. Serum creatinine < 2.0 mg/dL or calculated creatinine clearance (CrCl) > 45 mL/min
5. Patients must have adequate hepatic function obtained within 28 days prior to registration and documented by all of the following:

   * Total bilirubin ≤ 1.5 x IULN (≤ 5 x IULN if secondary to lymphoma, Gilbert's syndrome, or medication related)
   * Direct bilirubin ≤ 1.5 x IULN (≤ 5 x IULN if secondary to lymphoma)
   * AST and ALT ≤ 2.5 x IULN (≤ 5 x IULN secondary to lymphoma)
6. Patients must be willing to receive Pneumocystis jirovecii prophylaxis with sulfamethoxazole/trimethoprim, dapsone, and atovaquone or inhaled pentamadine, if they initiate combination umbralisib plus ublituximab (not for single agent ublituximab)
7. Patients must have a complete history and physical examination within 28 days prior to registration
8. Patients with follicular lymphoma must have the following components of Follicular Lymphoma International Prognostic Index (FLIPI) available from diagnosis, and collected again at time of registration:

   * Age
   * LDH
   * Number of nodal groups involved
   * Serum or plasma hemoglobin
   * Ann Arbor Stage Additionally, patients must have beta2-microglobulin collected at time of registration and response assessment.
9. Female subjects of reproductive potential must have a negative serum pregnancy test within 3 days prior to treatment start date. Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for ≥1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy at least six weeks ago) are exempt from pregnancy testing. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
10. Male and female subjects of reproductive potential who agree to use both a highly effective method of birth control (e.g., implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence, or sterilized partner) and a barrier method (e.g., condoms, cervical ring, sponge, etc.) during the period of therapy.

The following are UNACCEPTABLE forms of contraception for females of childbearing potential:

* natural family planning (rhythm method)
* breastfeeding
* fertility awareness
* withdrawal For subjects, these birth control requirements must be adhered to for 4 months after the last dose of umbralisib and 12 months after the last dose of ublituximab, whichever is later.

Regulatory Criteria

1. Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

Disease-Related

1. Transformed lymphoma; if clinical evidence of transformed lymphoma is present, transformation should be ruled out by biopsy of the suspicious lymph node/lesion
2. Prior treatment for follicular lymphoma or marginal zone lymphoma (Except: involved field or site radiation therapy is allowed)
3. Medically apparent central nervous system lymphoma or leptomeningeal disease
4. Tumor burden where administration of other FDA approved anti-CD20 antibodies like singleagent rituximab would be inappropriate.
5. Patients in need of immediate cytoreduction with chemotherapy based regimen.

Concurrent Conditions

1. Evidence of chronic active Hepatitis B (HBV, not including patients with prior hepatitis B vaccination; or positive serum Hepatitis B antibody) or chronic active Hepatitis C infection (HCV), active cytomegalovirus (CMV), or known history of HIV (or positive HIV test during screening). If HBc antibody is positive, the subject must be evaluated for the presence of HBV DNA by PCR. If HCV antibody is positive, the subject must be evaluated for the presence of HCV RNA by PCR. See Appendix: HEPATITIS B SEROLOGIC TEST RESULTS. If the subject is CMV IgG or CMV IgM positive, the subject must be evaluated for the presence of CMV DNA by PCR. Subjects with positive HBc antibody and negative HBV DNA by PCR are eligible. Subjects with positive HCV antibody and negative HCV RNA by PCR are eligible (subjects who are CMV IgG or CMV IgM positive but who are CMV DNA negative by PCR are eligible).
2. Ongoing drug-induced liver injury, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by stones, or cirrhosis of the liver
3. Inflammatory bowel disease (such as Crohn's disease or ulcerative colitis)
4. Irritable bowel syndrome with greater than 3 loose stools per day as a baseline
5. Active autoimmune disease requiring ongoing immunosuppressive therapy including systemic corticosteroids (prednisone or equivalent ≤10 mg daily allowed as clinically warranted) within 12 months prior to enrollment. Patients are allowed to use topical or inhaled corticosteroids or levothyroxine for hypothyroidism or hypogylcemic agents for diabetes mellitis.
6. Any severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study such as:

   * Symptomatic, or history of documented congestive heart failure NYHA (New York Heart Association) functional classification III-IV [see Appendix: New York Heart Association Classifications]
   * Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, CHF, or myocardial infarction within 6 months of enrollment.
   * Concomitant use of medication known to cause QT prolongation or torsades de pointes should be used with caution and at investigator discretion.
   * Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), angioplasty, cardiac or vascular stenting within 6 months of enrollment.
7. Women who are pregnant or lactating
8. History of other malignancies (including myelodysplastic syndromes) except:

   * malignancy treated with curative intent and with no known active disease present for >2 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician
   * adequately treated non-melanoma skin cancer without evidence of disease
   * adequately treated carcinoma in situ without evidence of disease
   * localized prostate cancer and PSA <1.0 mg/dL on 2 consecutive measurements at least 3 months apart with the most recent one being within 4 weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manali Kamdar, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gribben JG. How I treat indolent lymphoma. Blood. 2007 Jun 1;109(11):4617-26. doi: 10.1182/blood-2006-10-041863. Epub 2007 Feb 20. PMID 17311989
- [Background] Kahl BS. Follicular lymphoma: are we ready for a risk-adapted approach? Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):358-364. doi: 10.1182/asheducation-2017.1.358. PMID 29222279
- [Background] Relander T, Johnson NA, Farinha P, Connors JM, Sehn LH, Gascoyne RD. Prognostic factors in follicular lymphoma. J Clin Oncol. 2010 Jun 10;28(17):2902-13. doi: 10.1200/JCO.2009.26.1693. Epub 2010 Apr 12. PMID 20385990
- [Background] Campo E, Swerdlow SH, Harris NL, Pileri S, Stein H, Jaffe ES. The 2008 WHO classification of lymphoid neoplasms and beyond: evolving concepts and practical applications. Blood. 2011 May 12;117(19):5019-32. doi: 10.1182/blood-2011-01-293050. Epub 2011 Feb 7. PMID 21300984
- [Background] Horn H, Schmelter C, Leich E, Salaverria I, Katzenberger T, Ott MM, Kalla J, Romero M, Siebert R, Rosenwald A, Ott G. Follicular lymphoma grade 3B is a distinct neoplasm according to cytogenetic and immunohistochemical profiles. Haematologica. 2011 Sep;96(9):1327-34. doi: 10.3324/haematol.2011.042531. Epub 2011 Jun 9. PMID 21659362
- [Background] Link BK, Maurer MJ, Nowakowski GS, Ansell SM, Macon WR, Syrbu SI, Slager SL, Thompson CA, Inwards DJ, Johnston PB, Colgan JP, Witzig TE, Habermann TM, Cerhan JR. Rates and outcomes of follicular lymphoma transformation in the immunochemotherapy era: a report from the University of Iowa/MayoClinic Specialized Program of Research Excellence Molecular Epidemiology Resource. J Clin Oncol. 2013 Sep 10;31(26):3272-8. doi: 10.1200/JCO.2012.48.3990. Epub 2013 Jul 29. PMID 23897955
- [Background] Solal-Celigny P, Lepage E, Brousse N, Tendler CL, Brice P, Haioun C, Gabarre J, Pignon B, Tertian G, Bouabdallah R, Rossi JF, Doyen C, Coiffier B. Doxorubicin-containing regimen with or without interferon alfa-2b for advanced follicular lymphomas: final analysis of survival and toxicity in the Groupe d'Etude des Lymphomes Folliculaires 86 Trial. J Clin Oncol. 1998 Jul;16(7):2332-8. doi: 10.1200/JCO.1998.16.7.2332. PMID 9667247
- [Background] Solal-Celigny P. [Treatment of malignant low-grade lymphoma. Follicular Lymphoma Study Group]. Rev Med Interne. 1998;19 Suppl 1:18S-20S. doi: 10.1016/s0248-8663(98)80005-2. No abstract available. French. PMID 9789523
- [Background] Federico M, Bellei M, Marcheselli L, Luminari S, Lopez-Guillermo A, Vitolo U, Pro B, Pileri S, Pulsoni A, Soubeyran P, Cortelazzo S, Martinelli G, Martelli M, Rigacci L, Arcaini L, Di Raimondo F, Merli F, Sabattini E, McLaughlin P, Solal-Celigny P. Follicular lymphoma international prognostic index 2: a new prognostic index for follicular lymphoma developed by the international follicular lymphoma prognostic factor project. J Clin Oncol. 2009 Sep 20;27(27):4555-62. doi: 10.1200/JCO.2008.21.3991. Epub 2009 Aug 3. PMID 19652063
- [Background] Pastore A, Jurinovic V, Kridel R, Hoster E, Staiger AM, Szczepanowski M, Pott C, Kopp N, Murakami M, Horn H, Leich E, Moccia AA, Mottok A, Sunkavalli A, Van Hummelen P, Ducar M, Ennishi D, Shulha HP, Hother C, Connors JM, Sehn LH, Dreyling M, Neuberg D, Moller P, Feller AC, Hansmann ML, Stein H, Rosenwald A, Ott G, Klapper W, Unterhalt M, Hiddemann W, Gascoyne RD, Weinstock DM, Weigert O. Integration of gene mutations in risk prognostication for patients receiving first-line immunochemotherapy for follicular lymphoma: a retrospective analysis of a prospective clinical trial and validation in a population-based registry. Lancet Oncol. 2015 Sep;16(9):1111-1122. doi: 10.1016/S1470-2045(15)00169-2. Epub 2015 Aug 6. PMID 26256760
- [Background] Friedberg JW, Taylor MD, Cerhan JR, Flowers CR, Dillon H, Farber CM, Rogers ES, Hainsworth JD, Wong EK, Vose JM, Zelenetz AD, Link BK. Follicular lymphoma in the United States: first report of the national LymphoCare study. J Clin Oncol. 2009 Mar 10;27(8):1202-8. doi: 10.1200/JCO.2008.18.1495. Epub 2009 Feb 9. PMID 19204203
- [Background] Horning SJ, Rosenberg SA. The natural history of initially untreated low-grade non-Hodgkin's lymphomas. N Engl J Med. 1984 Dec 6;311(23):1471-5. doi: 10.1056/NEJM198412063112303. PMID 6548796
- [Background] Kahl BS, Hong F, Williams ME, Gascoyne RD, Wagner LI, Krauss JC, Habermann TM, Swinnen LJ, Schuster SJ, Peterson CG, Sborov MD, Martin SE, Weiss M, Ehmann WC, Horning SJ. Rituximab extended schedule or re-treatment trial for low-tumor burden follicular lymphoma: eastern cooperative oncology group protocol e4402. J Clin Oncol. 2014 Oct 1;32(28):3096-102. doi: 10.1200/JCO.2014.56.5853. Epub 2014 Aug 25. PMID 25154829
- [Background] Morschhauser F, Fowler NH, Feugier P, Bouabdallah R, Tilly H, Palomba ML, Fruchart C, Libby EN, Casasnovas RO, Flinn IW, Haioun C, Maisonneuve H, Ysebaert L, Bartlett NL, Bouabdallah K, Brice P, Ribrag V, Daguindau N, Le Gouill S, Pica GM, Martin Garcia-Sancho A, Lopez-Guillermo A, Larouche JF, Ando K, Gomes da Silva M, Andre M, Zachee P, Sehn LH, Tobinai K, Cartron G, Liu D, Wang J, Xerri L, Salles GA; RELEVANCE Trial Investigators. Rituximab plus Lenalidomide in Advanced Untreated Follicular Lymphoma. N Engl J Med. 2018 Sep 6;379(10):934-947. doi: 10.1056/NEJMoa1805104. PMID 30184451
- [Background] Rummel MJ, Niederle N, Maschmeyer G, Banat GA, von Grunhagen U, Losem C, Kofahl-Krause D, Heil G, Welslau M, Balser C, Kaiser U, Weidmann E, Durk H, Ballo H, Stauch M, Roller F, Barth J, Hoelzer D, Hinke A, Brugger W; Study group indolent Lymphomas (StiL). Bendamustine plus rituximab versus CHOP plus rituximab as first-line treatment for patients with indolent and mantle-cell lymphomas: an open-label, multicentre, randomised, phase 3 non-inferiority trial. Lancet. 2013 Apr 6;381(9873):1203-10. doi: 10.1016/S0140-6736(12)61763-2. Epub 2013 Feb 20. PMID 23433739
- [Background] Salles G, Seymour JF, Offner F, Lopez-Guillermo A, Belada D, Xerri L, Feugier P, Bouabdallah R, Catalano JV, Brice P, Caballero D, Haioun C, Pedersen LM, Delmer A, Simpson D, Leppa S, Soubeyran P, Hagenbeek A, Casasnovas O, Intragumtornchai T, Ferme C, da Silva MG, Sebban C, Lister A, Estell JA, Milone G, Sonet A, Mendila M, Coiffier B, Tilly H. Rituximab maintenance for 2 years in patients with high tumour burden follicular lymphoma responding to rituximab plus chemotherapy (PRIMA): a phase 3, randomised controlled trial. Lancet. 2011 Jan 1;377(9759):42-51. doi: 10.1016/S0140-6736(10)62175-7. Epub 2010 Dec 20. PMID 21176949
- [Background] Johnson PW, Rohatiner AZ, Whelan JS, Price CG, Love S, Lim J, Matthews J, Norton AJ, Amess JA, Lister TA. Patterns of survival in patients with recurrent follicular lymphoma: a 20-year study from a single center. J Clin Oncol. 1995 Jan;13(1):140-7. doi: 10.1200/JCO.1995.13.1.140. PMID 7799014
- [Background] Fisher RI, LeBlanc M, Press OW, Maloney DG, Unger JM, Miller TP. New treatment options have changed the survival of patients with follicular lymphoma. J Clin Oncol. 2005 Nov 20;23(33):8447-52. doi: 10.1200/JCO.2005.03.1674. Epub 2005 Oct 17. PMID 16230674
- [Background] Swenson WT, Wooldridge JE, Lynch CF, Forman-Hoffman VL, Chrischilles E, Link BK. Improved survival of follicular lymphoma patients in the United States. J Clin Oncol. 2005 Aug 1;23(22):5019-26. doi: 10.1200/JCO.2005.04.503. Epub 2005 Jun 27. PMID 15983392
- [Background] Armitage JO, Longo DL. Is watch and wait still acceptable for patients with low-grade follicular lymphoma? Blood. 2016 Jun 9;127(23):2804-8. doi: 10.1182/blood-2015-11-632745. Epub 2016 Mar 18. PMID 26994147
- [Background] Maddocks K, Barr PM, Cheson BD, Little RF, Baizer L, Kahl BS, Leonard JP, Fowler N, Gordon LI, Link BK, Friedberg JW, Ansell SM. Recommendations for Clinical Trial Development in Follicular Lymphoma. J Natl Cancer Inst. 2016 Dec 31;109(3):djw255. doi: 10.1093/jnci/djw255. Print 2017 Mar. PMID 28040699
- [Background] Kamdar MK, Smith SM. Extranodal Marginal Zone Lymphoma: No Longer Just a Sidekick. J Clin Oncol. 2017 Jun 10;35(17):1872-1878. doi: 10.1200/JCO.2017.72.2835. Epub 2017 Apr 27. PMID 28448239
- [Background] Thieblemont C. Improved biological insight and influence on management in indolent lymphoma. Talk 3: update on nodal and splenic marginal zone lymphoma. Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):371-378. doi: 10.1182/asheducation-2017.1.371. PMID 29222281
- [Background] Ardeshna KM, Qian W, Smith P, Braganca N, Lowry L, Patrick P, Warden J, Stevens L, Pocock CF, Miall F, Cunningham D, Davies J, Jack A, Stephens R, Walewski J, Ferhanoglu B, Bradstock K, Linch DC. Rituximab versus a watch-and-wait approach in patients with advanced-stage, asymptomatic, non-bulky follicular lymphoma: an open-label randomised phase 3 trial. Lancet Oncol. 2014 Apr;15(4):424-35. doi: 10.1016/S1470-2045(14)70027-0. Epub 2014 Mar 4. PMID 24602760
- [Background] Williams ME, Hong F, Gascoyne RD, Wagner LI, Krauss JC, Habermann TM, Swinnen LJ, Schuster SJ, Peterson CG, Sborov MD, Martin SE, Weiss M, Ehmann WC, Horning SJ, Kahl BS. Rituximab extended schedule or retreatment trial for low tumour burden non-follicular indolent B-cell non-Hodgkin lymphomas: Eastern Cooperative Oncology Group Protocol E4402. Br J Haematol. 2016 Jun;173(6):867-75. doi: 10.1111/bjh.14007. Epub 2016 Mar 11. PMID 26970533
- [Background] Conconi A, Martinelli G, Thieblemont C, Ferreri AJ, Devizzi L, Peccatori F, Ponzoni M, Pedrinis E, Dell'Oro S, Pruneri G, Filipazzi V, Dietrich PY, Gianni AM, Coiffier B, Cavalli F, Zucca E. Clinical activity of rituximab in extranodal marginal zone B-cell lymphoma of MALT type. Blood. 2003 Oct 15;102(8):2741-5. doi: 10.1182/blood-2002-11-3496. Epub 2003 Jul 3. PMID 12842999
- [Background] Kalpadakis C, Pangalis GA, Angelopoulou MK, Vassilakopoulos TP. Treatment of splenic marginal zone lymphoma. Best Pract Res Clin Haematol. 2017 Mar-Jun;30(1-2):139-148. doi: 10.1016/j.beha.2016.07.004. Epub 2016 Nov 4. PMID 28288709
- [Background] Sawas A, Farber CM, Schreeder MT, Khalil MY, Mahadevan D, Deng C, Amengual JE, Nikolinakos PG, Kolesar JM, Kuhn JG, Sportelli P, Miskin HP, O'Connor OA. A phase 1/2 trial of ublituximab, a novel anti-CD20 monoclonal antibody, in patients with B-cell non-Hodgkin lymphoma or chronic lymphocytic leukaemia previously exposed to rituximab. Br J Haematol. 2017 Apr;177(2):243-253. doi: 10.1111/bjh.14534. Epub 2017 Feb 21. PMID 28220479
- [Background] Mato AR, Shah NN, Jurczak W, Cheah CY, Pagel JM, Woyach JA, Fakhri B, Eyre TA, Lamanna N, Patel MR, Alencar A, Lech-Maranda E, Wierda WG, Coombs CC, Gerson JN, Ghia P, Le Gouill S, Lewis DJ, Sundaram S, Cohen JB, Flinn IW, Tam CS, Barve MA, Kuss B, Taylor J, Abdel-Wahab O, Schuster SJ, Palomba ML, Lewis KL, Roeker LE, Davids MS, Tan XN, Fenske TS, Wallin J, Tsai DE, Ku NC, Zhu E, Chen J, Yin M, Nair B, Ebata K, Marella N, Brown JR, Wang M. Pirtobrutinib in relapsed or refractory B-cell malignancies (BRUIN): a phase 1/2 study. Lancet. 2021 Mar 6;397(10277):892-901. doi: 10.1016/S0140-6736(21)00224-5. PMID 33676628
- [Background] Lannutti BJ, Meadows SA, Herman SE, Kashishian A, Steiner B, Johnson AJ, Byrd JC, Tyner JW, Loriaux MM, Deininger M, Druker BJ, Puri KD, Ulrich RG, Giese NA. CAL-101, a p110delta selective phosphatidylinositol-3-kinase inhibitor for the treatment of B-cell malignancies, inhibits PI3K signaling and cellular viability. Blood. 2011 Jan 13;117(2):591-4. doi: 10.1182/blood-2010-03-275305. Epub 2010 Oct 19. PMID 20959606
- [Background] Gopal AK, Kahl BS, de Vos S, Wagner-Johnston ND, Schuster SJ, Jurczak WJ, Flinn IW, Flowers CR, Martin P, Viardot A, Blum KA, Goy AH, Davies AJ, Zinzani PL, Dreyling M, Johnson D, Miller LL, Holes L, Li D, Dansey RD, Godfrey WR, Salles GA. PI3Kdelta inhibition by idelalisib in patients with relapsed indolent lymphoma. N Engl J Med. 2014 Mar 13;370(11):1008-18. doi: 10.1056/NEJMoa1314583. Epub 2014 Jan 22. PMID 24450858
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Lunning MA, Vose JM, Schreeder MT, et al: Ublituximab, a novel glycoengineered anti-CD20 mAb, in combination with TGR-1202, a next generation once daily PI3Kdelta inhibitor, demonstrates activity in heavily pretreated and high-risk chronic lymphocytic leukemia and B-cell lymphoma, American Society of Hematology. San Francisco, CA, 2014

RESULTS

PARTICIPANT FLOW:
Groups:
- Ublituximab Only: Treatment-Naive Stage II (non-contiguous), Stage III, Stage IV FL + MZL will receive Ublituximab 900mg IV weekly x 4 doses. End of treatment assessment 8 weeks post last dose of single agent ublituximab will be performed.
  During ublituximab monotherapy (initial treatment), Cycle 1 Day 1 administration time frame: Over 4 hours. Cycle 1 days 8 and 15 will be over 3 hours, and Cycle 1 Day 22 will be over 90 minutes.
- Ublituximab First, Then Ublituximab and Umbralisib: Patients who achieve less than a complete response will receive a combination of ublituximab and umbralisib for a total of 12 cycles. (In the combination arm ublituximab will be administered on day 1, 8, and 15 on cycle 1 and on day 1 on each cycle thereafter. Umbralisib will be administered at 800 mg daily for 12 cycles.
  During combination treatment with umbralisib, ublituximab will be administered over 90 minutes.
  Umbralisib will be administered orally once daily within 30 minutes of starting a meal.
Period: Cycle 1: Baseline to 8 Weeks
Arm/Group | Ublituximab Only | Ublituximab First, Then Ublituximab and Umbralisib
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0
Period: Cycle 2: 8 Weeks to 12 Months
Arm/Group | Ublituximab Only | Ublituximab First, Then Ublituximab and Umbralisib
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Ublituximab: Treatment-Naive Stage II (non-contiguous), Stage III, Stage IV FL + MZL will receive Ublituximab 900mg IV weekly x 4 doses. End of treatment assessment 8 weeks post last dose of single agent ublituximab will be performed. administered at 800 mg daily for 12 cycles)
- Experimental: Ublituximab and Umbralisib: Patients who achieve less than a complete response will receive a combination of ublituximab AND umbralisib for a total of 12 cycles. (In the combination arm ublituximab will be administered on day 1, 8, and 15 on cycle 1 and on day 1 on each cycle thereafter. Umbralisib will be administered at 800mg daily for 12 cycles)
- Total: Total of all reporting groups
Arm/Group | Experimental: Ublituximab | Experimental: Ublituximab and Umbralisib | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (6.3) | 66 (5.6) | 60.75 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response Rate (CR) at 8 Weeks Post Single Agent Induction
Description: Number of subjects that reached a complete response at the end of single agent induction as defined by a Lugano score of 3 or less on arm MONO - Monotherapy: Ublituximab.
  Complete response assessed via PET CT scan utilizing the Lugano-Deauville Criteria where none of the lymphoma lesions had FDG ( FluoroDeoxyglucose) avidity greater than the liver uptake.
  Patients who did not reach complete response at this point were then bridged to arm COMBO - Combotherapy: Ublituximab + Umbralisib.
Time Frame: 8 weeks post induction
Measure: Count of Participants; unit: Participants
Groups:
- Ublituximab Only: Monotherapy: Ublituximab
Arm/Group | Ublituximab Only
Number analyzed (Participants) | 4
Participants | 2

2. Primary Outcome: Number of Participants With Complete Response Rate (CR) at up to 12 Months Post MONO - Monotherapy: Ublituximab or Combotherapy: Ublituximab + Umbralisib.
Description: Number of subjects that reached a complete response at up to 12 months post induction as defined by a Lugano score of 3 or less on arms MONO - Monotherapy: Ublituximab.OR Combotherapy: Ublituximab + Umbralisib.
  Complete response assessed via PET CT scan utilizing the Lugano-Deauville Criteria where none of the lymphoma lesions had FDG ( FluoroDeoxyglucose) avidity greater than the liver uptake.
Time Frame: up to 12 months post induction
Measure: Count of Participants; unit: Participants
Groups:
- Ublituximab Only: Treatment-Naive Stage II (non-contiguous), Stage III, Stage IV FL + MZL will receive Ublituximab 900mg IV weekly x 4 doses. End of treatment assessment 8 weeks post last dose of single agent ublituximab will be performed.
  Ublituximab: Ublituximab will be administered as an intravenous infusion through a dedicated line. All infusions will be administered per institutional guidelines.
  During ublituximab monotherapy (initial treatment), Cycle 1 Day 1 administration time frame: Over 4 hours. Cycle 1 days 8 and 15 will be over 3 hours, and Cycle 1 Day 22 will be over 90 minutes. During combination treatment with umbralisib, ublituximab will be administered over 90 minutes.
- Ublituximab First, Then Ublituximab and Umbralisib: Patients who achieve less than a complete response on monotherapy Ublituximab will receive a combination of ublituximab AND umbralisib for a total of 12 cycles. (In the combination arm ublituximab will be administered on day 1,8 and 15 on cycle 1 and on day 1 on each cycle thereafter. Umbralisib will be administered at 800 mg daily for 12 cycles)
  Ublituximab: Ublituximab will be administered as an intravenous infusion through a dedicated line. All infusions will be administered per institutional guidelines.
  During ublituximab monotherapy (initial treatment), Cycle 1 Day 1 administration time frame: Over 4 hours. Cycle 1 days 8 and 15 will be over 3 hours, and Cycle 1 Day 22 will be over 90 minutes. During combination treatment with umbralisib, ublituximab will be administered over 90 minutes.
  Umbralisib: Umbralisib will be administered orally once daily within 30 minutes of starting a meal.
Arm/Group | Ublituximab Only | Ublituximab First, Then Ublituximab and Umbralisib
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

3. Secondary Outcome: Overall Response Rates (ORR) for Number of Participants
Description: Overall Response Rate for number of subjects as defined by a Lugano score of 3 or less on arms MONO - Monotherapy: Ublituximab.OR Combotherapy: Ublituximab + Umbralisib.
  Overall response rate assessed via PET CT utilizing Lugano deauvile criteria where lymphoma lesions had responded and would include complete response, partial response (> 50% improvement) and stable disease (less than 50 % response)
Time Frame: up to 12 months post induction
Measure: Count of Participants; unit: Participants
Arm/Group | Ublituximab Only | Ublituximab First, Then Ublituximab and Umbralisib
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: 15 months, 9 days
Groups:
- Ublituximab Only: Treatment-Naive Stage II (non-contiguous), Stage III, Stage IV FL + MZL will receive Ublituximab 900mg IV weekly x 4 doses. End of treatment assessment 8 weeks post last dose of single agent ublituximab will be performed.
  Ublituximab: Ublituximab will be administered as an intravenous infusion through a dedicated line. All infusions will be administered per institutional guidelines.
  During ublituximab monotherapy (initial treatment), Cycle 1 Day 1 administration time frame: Over 4 hours. Cycle 1 days 8 and 15 will be over 3 hours, and Cycle 1 Day 22 will be over 90 minutes.
- Ublituximab First, Then Ublituximab and Umbralisib: Patients who achieve less than a complete response will receive a combination of ublituximab AND umbralisib for a total of 12 cycles. (In the combination arm ublituximab will be administered on day 1,8 and 15 on cycle 1 and on day 1 on each cycle thereafter. Umbralisib will be administered at 800 mg daily for 12 cycles)
  During combination treatment with umbralisib, ublituximab will be administered over 90 minutes.
  Umbralisib: Umbralisib will be administered orally once daily within 30 minutes of starting a meal.
Arm/Group | Ublituximab Only | Ublituximab First, Then Ublituximab and Umbralisib
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ublituximab Only (N=2) | Ublituximab First, Then Ublituximab and Umbralisib (N=2)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Back Pain (General disorders) | 0 (0) | 1 (1)
volare bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Issues (Cardiac disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Visual Disturbance (Eye disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Mouth Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Elevated Transaminases (Hepatobiliary disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Nausea (General disorders) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Bilateral kidney pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Spasticity (Nervous system disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vaginal Infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT04508647/Prot_SAP_ICF_000.pdf